CLINICAL TRIAL: NCT01721785
Title: Diagnostic Value of Novel MR Imaging Techniques for the Primary Staging and Restaging of Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: 12-2-051; 2012-002935-27 (EudraCT Number)
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Rectal Neoplasms; Magnetic Resonance Imaging; Neoplasms Staging
Keywords: Nodal imaging; Restaging
MeSH Terms: conditions — Rectal Neoplasms | interventions — gadofosveset trisodium; Injections, Intravenous; Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary staging group I: All patients will be treated according to standard practice of the concerning hospital.
  Patients in group I are patients that will be stratified for direct surgery (TME) or a short-course of radiotherapy (5x5 Gy) followed by immediate TME.
  Group I will undergo only a staging MRI, including gadofosveset-enhanced MRI.
  Interventions: Drug: GADOFOSVESET TRISODIUM 244 Mg in 1 mL INTRAVENOUS INJECTION, SOLUTION [Ablavar]
- Restaging group II: All patients will be treated according to standard practice of the concerning hospital.
  Patients in group II are patients that will be stratified for a long course of chemoradiotherapy.
  Group II will undergo a staging MRI, a re-staging MRI and a optional sigmoidoscopy as part of restaging. MRI includes diffusion-weighted imaging and gadofosveset-enhanced MRI.
  Interventions: Drug: GADOFOSVESET TRISODIUM 244 Mg in 1 mL INTRAVENOUS INJECTION, SOLUTION [Ablavar]

INTERVENTIONS:
Drug: GADOFOSVESET TRISODIUM 244 Mg in 1 mL INTRAVENOUS INJECTION, SOLUTION [Ablavar] — Gadofosveset will be used as a lymph-node specific MRI contrast agent and will be administered by manual injection as a single intravenous bolus during MRI.
  Other Names: Ablavar; MS-325

SUMMARY:
The purpose of this study is to determine the clinical value of the novel MRI-techniques DWI and gadofosveset-enhanced MRI for the management of rectal cancer patients.

DETAILED DESCRIPTION:
Rectal cancer is a common form of cancer, and the treatment stratification depends on tumour and nodal stage as determined on MRI. Unfortunately, the information provided by standard T2-weighted MRI is not sufficient to accurately assess nodal involvement and tumour response after neo-adjuvant chemoradiotherapy. Additional functional information is required for reliable (re)staging. Diffusion-weighted imaging and gadofosveset-enhanced MRI are two new imaging techniques that have all shown great potential in rectal cancer staging. In order to provide definite evidence there is a need for a multicenter study with a large patient population.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven primary rectal cancer (≤15 cm from the anorectal verge as measured in MRI)
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Ineligibility to undergo MRI (claustrophobia, pacemaker, non-MR compatible surgical implants, metal fragments in the eye)
* Pregnancy
* Locally recurrent rectal cancer
* A history of severe allergy to contrast agents
* Ineligibility to receive gadofosveset contrast (history of contrast allergy, impaired kidney function with a Glomerular Filtration Rate <30 ml/min/1.73m2
* Incurable disease due to metastases or co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with rectal cancer in one of the participating centres will be considered for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2012-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the techniques under investigation | 2 years
  Techniques under investigation are diffusion-weighted imaging for tumour response assessment and gadofosveset-enhanced MRI for nodal assessment, compared to standard T2-weighted MRI.

SECONDARY OUTCOMES:
To determine the inter-observer agreement for the imaging techniques under investigation | 2 years
  Detection of the differences between expert vs non-expert readers and general vs referral centres concerning diffusion-weighted imaging and gadofosveset-enhanced MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Beets-Tan, Prof. MD., Principal Investigator — Radiology, MUMC; Geerard Beets, Ass Prof. MD, Principal Investigator — Surgery, MUMC; Doenja Lambregts, MD, Study Chair — Radiology, MUMC; Monique Maas, MD, Study Chair — Radiology, MUMC
Locations (10):
- Netherlands (10):
  - Atrium Medisch Centrum, Heerlen, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg
  - Orbis Medisch Centrum, Sittard-Geleen, Limburg
  - Viecuri Medisch Centrum, Venlo, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Amphia Ziekenhuis, Breda, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - AMC, Amsterdam, North Holland
  - ZGT, Almelo, Overrijsel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lahaye MJ, Engelen SM, Nelemans PJ, Beets GL, van de Velde CJ, van Engelshoven JM, Beets-Tan RG. Imaging for predicting the risk factors--the circumferential resection margin and nodal disease--of local recurrence in rectal cancer: a meta-analysis. Semin Ultrasound CT MR. 2005 Aug;26(4):259-68. doi: 10.1053/j.sult.2005.04.005. PMID 16152740
- [Background] Maas M, Beets-Tan RG, Lambregts DM, Lammering G, Nelemans PJ, Engelen SM, van Dam RM, Jansen RL, Sosef M, Leijtens JW, Hulsewe KW, Buijsen J, Beets GL. Wait-and-see policy for clinical complete responders after chemoradiation for rectal cancer. J Clin Oncol. 2011 Dec 10;29(35):4633-40. doi: 10.1200/JCO.2011.37.7176. Epub 2011 Nov 7. PMID 22067400
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Background] Lambregts DM, Beets GL, Maas M, Kessels AG, Bakers FC, Cappendijk VC, Engelen SM, Lahaye MJ, de Bruine AP, Lammering G, Leiner T, Verwoerd JL, Wildberger JE, Beets-Tan RG. Accuracy of gadofosveset-enhanced MRI for nodal staging and restaging in rectal cancer. Ann Surg. 2011 Mar;253(3):539-45. doi: 10.1097/SLA.0b013e31820b01f1. PMID 21239980
- [Background] Herborn CU, Lauenstein TC, Vogt FM, Lauffer RB, Debatin JF, Ruehm SG. Interstitial MR lymphography with MS-325: characterization of normal and tumor-invaded lymph nodes in a rabbit model. AJR Am J Roentgenol. 2002 Dec;179(6):1567-72. doi: 10.2214/ajr.179.6.1791567. PMID 12438057
- [Background] Yamashita T, Takahara T, Kwee TC, Kawada S, Horie T, Inomoto C, Hashida K, Yamamuro H, Myojin K, Luijten PR, Imai Y. Diffusion magnetic resonance imaging with gadofosveset trisodium as a negative contrast agent for lymph node metastases assessment. Jpn J Radiol. 2011 Jan;29(1):25-32. doi: 10.1007/s11604-010-0513-2. Epub 2011 Jan 26. PMID 21264658
- [Background] Kim SH, Lee JY, Lee JM, Han JK, Choi BI. Apparent diffusion coefficient for evaluating tumour response to neoadjuvant chemoradiation therapy for locally advanced rectal cancer. Eur Radiol. 2011 May;21(5):987-95. doi: 10.1007/s00330-010-1989-y. Epub 2010 Oct 27. PMID 20978768
- [Background] Kim SH, Lee JM, Hong SH, Kim GH, Lee JY, Han JK, Choi BI. Locally advanced rectal cancer: added value of diffusion-weighted MR imaging in the evaluation of tumor response to neoadjuvant chemo- and radiation therapy. Radiology. 2009 Oct;253(1):116-25. doi: 10.1148/radiol.2532090027. PMID 19789256
- [Background] Lambregts DM, Vandecaveye V, Barbaro B, Bakers FC, Lambrecht M, Maas M, Haustermans K, Valentini V, Beets GL, Beets-Tan RG. Diffusion-weighted MRI for selection of complete responders after chemoradiation for locally advanced rectal cancer: a multicenter study. Ann Surg Oncol. 2011 Aug;18(8):2224-31. doi: 10.1245/s10434-011-1607-5. Epub 2011 Feb 23. PMID 21347783
- [Background] Curvo-Semedo L, Lambregts DM, Maas M, Thywissen T, Mehsen RT, Lammering G, Beets GL, Caseiro-Alves F, Beets-Tan RG. Rectal cancer: assessment of complete response to preoperative combined radiation therapy with chemotherapy--conventional MR volumetry versus diffusion-weighted MR imaging. Radiology. 2011 Sep;260(3):734-43. doi: 10.1148/radiol.11102467. Epub 2011 Jun 14. PMID 21673229
- [Background] Habr-Gama A, Perez RO, Wynn G, Marks J, Kessler H, Gama-Rodrigues J. Complete clinical response after neoadjuvant chemoradiation therapy for distal rectal cancer: characterization of clinical and endoscopic findings for standardization. Dis Colon Rectum. 2010 Dec;53(12):1692-8. doi: 10.1007/DCR.0b013e3181f42b89. PMID 21178866